CLINICAL TRIAL: NCT02075801
Title: Longitudinal Results of a 10-years Clinical Trial of Sealed Margin Failures of Amalgam Restorations
Brief Title: 10-years Clinical Trial of Sealed of Margin Failures
Acronym: Sealant
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Gustavo Moncada, Main Investigator, University of Chile
Other Study IDs: PRI-ODO-0207
Record Dates: First submitted 2014-02-21; First posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Dental Caries Secondary to Acquired Defects of Tooth Structure
Keywords: Sealant, Margins Defect, Amalgam

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Defective amalgam restorations: Treatment Groups:
  A. Sealing of amalgam margin defects: Defective areas were acid etched with 35% phosphoric acid for 15 seconds. A resin-based sealant (Sealant, 3MESPE)was applied over the defective area. The sealant was polymerized with a photo curing unit (Curing-Light 2500, 3MESPE) for 40 seconds. Rubber dam isolation was used for this procedure. All treatments were applied by the same clinician.
  B. Replacement Group: The clinician totally removed and replaces the defective restoration with a new amalgam (Tytin, Kerr, Orange, USA). Rubber dam isolation was used for this procedure. All treatments were applied by the same clinician.
  C. Control Group: The defective restorations did not receive any treatment.
  Interventions: Other: Sealing of amalgam margin defects

INTERVENTIONS:
Other: Sealing of amalgam margin defects — Comparison between sealing of amalgam margins defects, replacement and non treated groups.
Other: Sealing of amalgam margin defects — A.Sealing of amalgam margin defects: were acid etched with 35% phosphoric acid for 15 seconds. A resin-based sealant (Clinpro Sealant, 3MESPE) was applied over the defective area. The sealant was polymerized with a photocuring unit (Curing Light 2500, 3M ESPE) for 40 seconds. Rubber dam isolation was used for this procedure. All treatments were applied by the same clinician.
  B.Replacement Group: The clinician totally removed and replaces the defective restoration with a new amalgam (Tytin, Kerr Corporation, Orange, CA, USA). Rubber dam isolation was used for this procedure. All treatments were applied by the same clinician.
  C.Control Group: The defective restorations did not receive any treatment.
  Other Names: Use of Selant to seal amalgam margins defects

SUMMARY:
* Assess the effectiveness of sealing localized marginal defects of amalgam restorations that were initially scheduled for replacement of restorations.
* The hypothesis was that sealed defective margins of the amalgam restorations shows similar performance than replacement amalgam restorations.

DETAILED DESCRIPTION:
Study Design

Were examined 157 patients with 586 amalgam restorations that were recruited at the Operative Dentistry Clinic, at the Dental School, University of Chile with the indication of amalgam replacements, of them, a cohort of thirty two patients (19 females and 13 males, mean age = 27 years old), with 73 Class I amalgam restorations, that presented one or more localized margin defects (Bravo or Charlie according to modified United State Public Health Service, USPHS criteria), were included in the study. The protocol was approved by the Institutional Research Ethics Committee of the Dental School at the University of Chile, Investigation Project, School of Dentistry (0205) and all patients signed the informed consent form and completed the registration form. Only Faculty members were accepted to provide the treatment.

Treatment Groups Criteria: 73 restorations with defective margins were evaluated in accordance with the modified USPHS criteria and assigned to either the sealant (n=26), repair (n=21) and control groups (n=26).

Restorations Assessment: The quality of the restorations were evaluated using the modified U.S. Public Health System/Ryge criteria. Two examiners assessed the restorations independently and by visual and tactile (mouth mirror number 5) examination using an explorer (N° 23) and indirectly by radiographic, examination, for interproximal observation (Bite Wing). All the restorations were examined at baseline and each year during four and ten years after treatment. The restorations assessment was carried out by five parameters: marginal adaptation (MA), roughness (R), secondary caries (SC), marginal stain (MS) and teeth sensitivity (TS). If any difference was recorded between the 2 independent examiners, and they did not reach an agreement, a third clinician was called to assist with the process decision. If the three clinicians they did not reach an agreement, the lower score was recorded. All three clinicians participated in calibration exercises at the beginning and before the last examination took place and the inter-examiner reliability results were Kappa=0.74 at the baseline and Kappa=0.87 at the ten year.

A change from Bravo to Alpha was considered an improvement and a change from Alpha to Bravo was considered downgrade.

Caries risk assessment: A graphical computed program (CARIOGRAM) was used for individual´s patients caries risk assessed, the program weighted the interaction between the following 10 caries related factors: Caries experience, related general disease, diet contents, diet frequency, plaque amount by Silness Löe Index, semi quantitative detection of mutans streptococci and lactobacilli in saliva by Caries Risk Test (CRT), fluoride program, amount of saliva stimulated secretion by CRT Buffer (Vivadent), saliva buffer capacity and clinical judgment. Patients were classifying in high, intermediate and low caries risk. Additionally the results also indicate where targeted actions to improve the situation will have the best effect.

Patients were recalled ten years after the treatment, for clinical assessment by the same examiners, applying the same criteria used at baseline. Failed restorations were removed from the study and treated according to the diagnosed needs.

Statistical analysis The ordinal dependent variable was changed in level of the modified USPHS criteria from the baseline value. The assigned score of each restoration reflected the worst result for any of the parameters. The results of each group in terms of degradation or upgrade were analyzed by Friedman range non-parametric test to compare the pre and postoperative conditions. Additionally, the performance of all groups was contrasted using the Mann Whitney test to determine the differences between the upgrade and downgrade of the restoration´s quality. The statistical significance was set at 95%, α=0.05 and β=0.80 for statistical analysis.

ELIGIBILITY:
Inclusion criteria:

* Patients with amalgam restorations with marginal deficiencies that were judged to be suitable for sealing.
* Older than 18 years of age ¨
* More than 20 teeth in their mouth
* The restorations had to be in functional occlusion with an opposing natural tooth
* With at least one proximal contact area with and adjacent tooth
* Area out of the restoration´s failures in good condition
* Patients who agree and sign the informed consent for participating in the study.

Exclusion Criteria:

* Patients with contraindications for regular dental treatment based on their medical history
* Special aesthetic requirements that could not be solved by this alternative treatment
* Xerostomia or who were taking medication that significantly decreased salivary flow
* High caries risk
* Psychiatric or physical diseases, that interfered with teeth hygiene.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of the Operative Dentistry Clinics, School of Dentistry, University of Chile
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2003-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Changes of Amalgam restorations quality according to United Stated Public Health Service (USPHS) | Baseline and 10 after treatment
  Restorations Assessment: The quality of the restorations were evaluated using the modified U.S. Public Health System criteria. Two examiners assessed the restorations independently and by visual and tactile examination. All the restorations were examined at baseline and ten years after treatment. The restorations assessment was carried out by five parameters: marginal adaptation, roughness, secondary caries, marginal stain and teeth sensitivity. All three clinicians participated in calibration exercises at the beginning and before the last examination took place and the inter-examiner reliability results were Kappa=0.74 at the baseline and Kappa=0.87 at the ten year.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Moncada, DDS, Principal Investigator — University of Chile
Locations (1):
- University of Chile, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Martin J, Fernandez E, Estay J, Gordan VV, Mjor IA, Moncada G. Management of Class I and Class II Amalgam Restorations with Localized Defects: Five-Year Results. Int J Dent. 2013;2013:450260. doi: 10.1155/2013/450260. Epub 2013 Jan 28. PMID 23431302
- [Background] Martin J, Fernandez E, Estay J, Gordan VV, Mjor IA, Moncada G. Minimal invasive treatment for defective restorations: five-year results using sealants. Oper Dent. 2013 Mar-Apr;38(2):125-33. doi: 10.2341/12-062C. Epub 2012 Jul 11. PMID 22788726
- [Background] Moncada G, Angel P, Fernandez E, Alonso P, Martin J, Gordan VV. Bond strength evaluation of nanohybrid resin-based composite repair. Gen Dent. 2012 May-Jun;60(3):230-4. PMID 22623463
- [Background] Fernandez EM, Martin JA, Angel PA, Mjor IA, Gordan VV, Moncada GA. Survival rate of sealed, refurbished and repaired defective restorations: 4-year follow-up. Braz Dent J. 2011;22(2):134-9. doi: 10.1590/s0103-64402011000200008. PMID 21537587
- [Background] Moncada G, Martin J, Fernandez E, Hempel MC, Mjor IA, Gordan VV. Sealing, refurbishment and repair of Class I and Class II defective restorations: a three-year clinical trial. J Am Dent Assoc. 2009 Apr;140(4):425-32. doi: 10.14219/jada.archive.2009.0191. PMID 19339531
- [Background] Moncada G, Fernandez E, Martin J, Arancibia C, Mjor IA, Gordan VV. Increasing the longevity of restorations by minimal intervention: a two-year clinical trial. Oper Dent. 2008 May-Jun;33(3):258-64. doi: 10.2341/07-113. PMID 18505215
- [Background] Moncada GC, Martin J, Fernandez E, Vildosola PG, Caamano C, Caro MJ, Mjor IA, Gordan VV. Alternative treatments for resin-based composite and amalgam restorations with marginal defects: a 12-month clinical trial. Gen Dent. 2006 Sep-Oct;54(5):314-8. PMID 17004564